CLINICAL TRIAL: NCT02313363
Title: Feasibility of a Patient-Centered Smartphone-Based Diabetes Care System: a Pilot Study
Brief Title: Patient-Centered Smartphone-Based Diabetes Care
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: H-1301-075-459
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Health care systems; Mobile applications; Self-care; Diabetes mellitus; Smartphone
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PSDCS (Experimental): using the patient-centered smartphone-based diabetes care system (PSDCS) for 12 weeks
  Interventions: Device: patient-centered smartphone-based diabetes care system

INTERVENTIONS:
Device: patient-centered smartphone-based diabetes care system — patient-centered smartphone-based diabetes care system (PSDCS) is composed of 4 modules such as glucose module, diet module, physical activity module, and SNS module. Participants were instructed to use the PSDCS and to measure blood glucose levels with a Bluetooth glucometer, input daily food intake, and wear an activity tracker.

SUMMARY:
The investigators developed a patient-centered smartphone-based diabetes care system (PSDCS). This study was aimed to test the feasibility of the PSDCS.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* HbA1c levels ≥ 6.5%

Exclusion Criteria:

* severe diabetic complication including severe non-proliferative diabetic retinopathy or proliferative diabetic retinopathy, chronic kidney disease stage 4-5, severe diabetic neuropathy, history of diabetic foot, history of angina pectoris, myocardial infarction, and cerebrovascular disease, and peripheral arterial disease
* type 1 diabetes
* insulin therapy other than insulin glargine
* subjects with insulin pump
* history of drug addiction
* history of psychotic disorder
* pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
change of HbA1c | baseline and the end of 12 week

SECONDARY OUTCOMES:
change of fasting plasma glucose | baseline and after 12 weeks (within 3 days)
change of lipid profile | baseline and after 12 weeks (within 3 days)
change of body weight | baseline and after 12 weeks (within 3 days)
change of the scores of Summary of Diabetes Self-Care Activities (SDSCA) | baseline and after 12 weeks (within 3 days)

OTHER OUTCOMES:
number of events of serious hyperglycemia | 12 weeks
  320 mg/dL or higher by the glucometer readouts
number of events of hypoglycemia | 12 weeks
  less than 70 mg/dL by the glucometer readouts

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PHD, Principal Investigator — Seoul National University Hospital